CLINICAL TRIAL: NCT00001481
Title: An Endocrine Model for Postpartum Mood Disorders
Brief Title: The Role of Hormones in Postpartum Mood Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 950097; 95-M-0097
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-01-15

CONDITIONS: Postpartum Depression
Keywords: Postpartum Disorders; Mood; Hormones; GnRH Agonist; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Estradiol; Progesterone; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1a - Postpartum depression: Hormone withdrawal Group (Experimental): Female participants with history of postpartum depression (PPD) received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 15, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily. During weeks 16 through 20, all participants received placebo capsules to be taken twice daily.
  Interventions: Drug: Estradiol; Other: Placebo; Drug: Progesterone; Drug: leuprolide acetate
- Arm 1b - Depression, non-reproductive: Hormone withdrawal Group (Experimental): Female participants with history of non-reproductive related depression received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 15, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily. During weeks 16 through 20, all participants received placebo capsules to be taken twice daily.
  Interventions: Drug: Estradiol; Other: Placebo; Drug: Progesterone; Drug: leuprolide acetate
- Arm 1c- Healthy Volunteer: Hormone withdrawal Group (Active Comparator): Female participants without history of depression received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 15, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily. During weeks 16 through 20, all participants received placebo capsules to be taken twice daily.
  Interventions: Drug: Estradiol; Other: Placebo; Drug: Progesterone; Drug: leuprolide acetate
- Arm 2a: Postpartum Depression; Hormone Continuation Group (Experimental): Female participants with history of postpartum depression (PPD) received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 20, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily.
  Interventions: Drug: Estradiol; Other: Placebo; Drug: Progesterone; Drug: leuprolide acetate
- Arm 2b - Depression, non-reproductive: Hormone Continuation Group (Experimental): Female participants with history of non-reproductive related depression received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 20, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily.
  Interventions: Drug: Estradiol; Other: Placebo; Drug: Progesterone; Drug: leuprolide acetate
- Arm 2c- Healthy Volunteer: Hormone Continuation Group (Active Comparator): Female participants without history of depression received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 20, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily.
  Interventions: Drug: Estradiol; Other: Placebo; Drug: Progesterone; Drug: leuprolide acetate

INTERVENTIONS:
Drug: Estradiol — Participants receive 17 beta-estradiol as oral capsule twice daily
Other: Placebo — Participants receive placebo as oral capsule twice daily
Drug: Progesterone — Participants receive progesterone as oral capsule twice daily
Drug: leuprolide acetate — Leuprolide acetate is a gonadotropin releasing hormone (GnRH) agonist, given via intramuscular injection monthly
  Other Names: Lupron

SUMMARY:
The present protocol is designed to create a "scaled-down" hormonal milieu of pregnancy and the puerperium in order to determine whether it is the abrupt withdrawal of gonadal steroids or the prolonged exposure to gonadal steroids that is associated with mood symptoms.

DETAILED DESCRIPTION:
The appearance of mood and behavioral symptoms during pregnancy and the postpartum period has been extensively reported. While there has been much speculation about possible biologically based etiologies for postpartum disorders (PPD), none has ever been confirmed. The present protocol is designed to create a "scaled-down" hormonal milieu of pregnancy and the puerperium in order to determine whether women who have had a previous episode of postpartum major affective episode will experience differential mood and behavioral effects during ovarian hormone exposure and/or withdrawal compared with controls and to determine whether it is the abrupt withdrawal of gonadal steroids or the prolonged exposure to gonadal steroids that is associated with mood symptoms. Supraphysiologic plasma levels of gonadal steroids will be established, maintained, and then rapidly reduced, simulating the hormonal events that occur during pregnancy and parturition. This will be accomplished by administering estradiol and progesterone to women who are pretreated with a gonadotropin releasing hormone (GnRH) agonist (Lupron). After eight weeks, administration of gonadal steroids will be stopped in one group of patients and controls, and a sudden decline in the plasma hormone levels will be precipitated. Another group will be maintained on supraphysiologic levels of estrogen and progesterone for an additional month.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Group 1: Women with a history of postpartum depression:

1. A history of Diagnostic and Statistical Manual (DSM)-IV major depression or hypomanic/manic episode that occurred within three months of childbirth (as determined by a Structured Clinical Interview for the DSM (SCID) interview));
2. has been well for a minimum of one year;
3. a regular menstrual cycle for at least three months;
4. age 18-50;
5. not pregnant, not lactating and in good medical health;
6. medication free (including birth control pills);
7. no history of puerperal suicide attempts or psychotic episodes requiring hospitalization.

B. Group 2: Women with a history of Major Depressive Disorder

1. A history of DSM-IV major depression episode(s) occurring outside of pregnancy and not within three months postpartum;
2. has been well for a minimum of one year;
3. a regular menstrual cycle for at least three months;
4. age 18-50;
5. not pregnant, not lactating and in good medical health;
6. medication free (including birth control pills);
7. no history of suicide attempts or psychotic episodes requiring hospitalization.

C. Group 3: Normal Controls

1) Controls will meet all criteria specified except they must not have any past or present Axis I diagnosis or evidence of menstrual related mood disorders.

EXCLUSION CRITERIA:

Patients will not be permitted to enter this protocol if they have important clinical or laboratory abnormalities including any history of the following:

* endometriosis;
* undiagnosed enlargement of the ovaries;
* liver disease;
* breast cancer;
* a history of blood clots in the legs or lungs;
* undiagnosed vaginal bleeding;
* porphyria;
* diabetes mellitus;
* malignant melanoma;
* gallbladder or pancreatic disease;
* heart or kidney disease;
* cerebrovascular disease (stroke);
* cigarette smoking;
* a history of suicide attempts or psychotic episodes requiring hospitalization;
* recurrent migraine headaches;
* pregnancy (patients will be warned not to become pregnant during the study and will be advised to employ barrier contraceptive methods;
* pregnancy-related medical conditions such as hyperemesis gravidarum, pretoxemia and toxemia, deep vein thrombosis (DVT) and bleeding diathesis;
* Any woman with a first degree relative (immediate family) with premenopausal breast cancer or breast cancer presenting in both breasts or any woman who has multiple family members (greater than three relatives) with postmenopausal breast cancer will also be excluded from participating in this protocol;
* Any woman meeting the Stages of Reproductive Aging Workshop Criteria (STRAW) for the perimenopause will be excluded from participation. Specifically, we will exclude any woman with an elevated plasma follicle stimulating hormone (FSH) level (greater than or equal to 14 IU/L) and with menstrual cycle variability of > 7 days different from their normal cycle length;
* Subjects who are unable to provide informed consent;
* National Institute of Mental Health (NIMH) employees and staff and their immediate family members will be excluded from the study per NIMH policy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 1996-04-26 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with dbGaP, BTRIS and NIMH Data Archive as determined by the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 24 months after final publication
Access Criteria: Data will be shared with dbGaP, Biomedical Translational Research Information System (BTRIS) and NIMH Data Archive as determined by the Principal Investigator.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1995-M-0097.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 74 participants were consented:
  * 21 participants were screen failure
  * 2 participants withdrew after signing consent
  * 4 participants dropped out prior to randomization
  * 1 participant dropped out after randomization and prior to start of intervention
  * 46 participants were randomized and received study intervention
Groups:
- Arm 1a - Postpartum Depression: Hormone Withdrawal: Female participants with history of postpartum depression (PPD) received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 15, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily. During weeks 16 through 20, all participants received placebo capsules to be taken twice daily.
- Arm 1b - Depression, Non-reproductive: Hormone Withdrawal: Female participants with history of non-reproductive related depression received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 15, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily. During weeks 16 through 20, all participants received placebo capsules to be taken twice daily.
- Arm 1c - Healthy Volunteer: Hormone Withdrawal: Female participants without history of depression received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 15, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily. During weeks 16 through 20, all participants received placebo capsules to be taken twice daily.
- Arm 2a - Postpartum Depression: Hormone Continuation: Female participants with history of postpartum depression (PPD) received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 20, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily.
- Arm 2b - Depression, Non-reproductive: Hormone Continuation: Female participants with history of non-reproductive related depression received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 20, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily.
- Arm 2c - Healthy Volunteer: Hormone Continuation: Female participants without history of depression received 3.75 mg of gonadotropin releasing hormone (GnRH) agonist leuprolide acetate (Lupron) via intramuscular injection on a monthly basis for five months (20 weeks), administered during visit for weeks 0, 4, 8, 12, & 16. Participants received oral capsules twice daily under single blind conditions for the same 5 months (20 weeks). During weeks 0 through 7, all participants received placebo via oral capsule twice daily. During weeks 8 through 20, all participants received 2 mg of 17 beta-estradiol via oral capsule twice daily and 200 mg of progesterone via oral capsule twice daily.
Period: Study 1
Arm/Group | Arm 1a - Postpartum Depression: Hormone Withdrawal | Arm 1b - Depression, Non-reproductive: Hormone Withdrawal | Arm 1c - Healthy Volunteer: Hormone Withdrawal | Arm 2a - Postpartum Depression: Hormone Continuation | Arm 2b - Depression, Non-reproductive: Hormone Continuation | Arm 2c - Healthy Volunteer: Hormone Continuation
Started | 7 | 0 | 8 | 0 | 0 | 0
Completed | 7 | 0 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Study 2
Arm/Group | Arm 1a - Postpartum Depression: Hormone Withdrawal | Arm 1b - Depression, Non-reproductive: Hormone Withdrawal | Arm 1c - Healthy Volunteer: Hormone Withdrawal | Arm 2a - Postpartum Depression: Hormone Continuation | Arm 2b - Depression, Non-reproductive: Hormone Continuation | Arm 2c - Healthy Volunteer: Hormone Continuation
Started | 9 | 1 | 5 | 7 | 2 | 7
Completed | 9 | 1 | 5 | 7 | 2 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1a - Postpartum Depression: Hormone Withdrawal Group | Arm 1b - Depression, Non-reproductive: Hormone Withdrawal Group | Arm 1c- Healthy Volunteer: Hormone Withdrawal Group | Arm 2a: Postpartum Depression; Hormone Continuation Group | Arm 2b - Depression, Non-reproductive: Hormone Continuation Group | Arm 2c- Healthy Volunteer: Hormone Continuation Group | Total
Number analyzed (Participants) | 16 | 1 | 13 | 7 | 2 | 7 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 0 | 2 | 0 | 0 | 5
  Between 18 and 65 years | 13 | 1 | 13 | 5 | 2 | 7 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 1 | 13 | 7 | 2 | 7 | 46
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 15 | 1 | 12 | 6 | 2 | 7 | 43
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 7 | 2 | 1 | 4 | 16
  White | 12 | 1 | 5 | 4 | 1 | 1 | 24
  More than one race | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Edinburgh Postnatal Depression Scale (EPDS) Mean Total Score
Description: The Edinburgh Postnatal Depression Scale (EPDS) is a self-reported 10 item questionnaire to asses a participant's mood over the past week. Each question has four possible answers, scored from 0 to 3 with total score ranging from 0 to 30. Higher scores indicate more severe mood symptoms. EPDS was administered once every 2 weeks for the duration of the study. Analysis was calculated as the mean of scores for baseline (week 16) and weeks 18 and 20.
Time Frame: Weeks 16, 18, and 20
Population: Analysis applies to participants in study 2. Two participants did not complete rating in week 16. One participant did not complete rating in week 18. Two participants did not complete rating in week 20.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1a - Postpartum Depression: Hormone Withdrawal | Arm 1b - Depression, Non-reproductive: Hormone Withdrawal | Arm 1c - Healthy Volunteer: Hormone Withdrawal | Arm 2a - Postpartum Depression: Hormone Continuation | Arm 2b - Depression, Non-reproductive: Hormone Continuation | Arm 2c - Healthy Volunteer: Hormone Continuation
Number analyzed (Participants) | 9 | 1 | 5 | 7 | 2 | 7
Units on a scale
  Week 16: number analyzed (Participants) | 8 | 1 | 5 | 7 | 2 | 6
  Week 16 | 3.75 (6.32) | 3 (NA) — Standard Deviation is not calculable for one participant | 0 (0) | 1.14 (1.07) | 0.5 (0.71) | 0.67 (1.21)
  Week 18: number analyzed (Participants) | 9 | 1 | 5 | 7 | 1 | 7
  Week 18 | 1.22 (3.31) | 0 (NA) — Standard Deviation is not calculable for one participant | 0 (0) | 2.29 (2.36) | 0 (NA) — Standard Deviation is not calculable for one participant | 0.29 (0.49)
  Week 20: number analyzed (Participants) | 8 | 1 | 5 | 7 | 2 | 6
  Week 20 | 1 (1.93) | 0 (NA) — Standard Deviation is not calculable for one participant | 0.2 (0.45) | 3.71 (4.54) | 0.5 (0.71) | 0.67 (0.82)

ADVERSE EVENTS:
Time Frame: Up to 28 weeks from start of study
Arm/Group | Arm 1a - Postpartum Depression: Hormone Withdrawal | Arm 1b - Depression, Non-reproductive: Hormone Withdrawal | Arm 1c - Healthy Volunteer: Hormone Withdrawal | Arm 2a - Postpartum Depression: Hormone Continuation | Arm 2b - Depression, Non-reproductive: Hormone Continuation | Arm 2c - Healthy Volunteer: Hormone Continuation
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/1 | 0/13 | 0/7 | 0/2 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/1 | 0/13 | 0/7 | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 3/16 | 0/1 | 0/13 | 1/7 | 0/2 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1a - Postpartum Depression: Hormone Withdrawal (N=16) | Arm 1b - Depression, Non-reproductive: Hormone Withdrawal (N=1) | Arm 1c - Healthy Volunteer: Hormone Withdrawal (N=13) | Arm 2a - Postpartum Depression: Hormone Continuation (N=7) | Arm 2b - Depression, Non-reproductive: Hormone Continuation (N=2) | Arm 2c - Healthy Volunteer: Hormone Continuation (N=7)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT00001481/Prot_SAP_000.pdf